CLINICAL TRIAL: NCT03923387
Title: A Multicenter, Open Label, Prospective, Randomized Study of the MynxGrip Vascular Closure Device in Subjects With Diagnostic or Interventional Endovascular Procedures (PANDA Study)
Brief Title: Study to Evaluate the Safety and Effectiveness of MynxGrip Vascular Closure Device
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17-0005
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2020-08

CONDITIONS: Endovascular
Keywords: Vascular closure

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel controlled trial, in which treatment is conducted simultaneously for both the test group and the control group, so that potential differences influencing the outcome measures between both groups can be minimized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MynxGrip (Experimental): MynxGrip, a vascular closure device indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F or 7F procedural sheath.
  Interventions: Device: MynxGrip
- Manual compression (Active Comparator): Manual compression hemostasis
  Interventions: Other: Manual compression

INTERVENTIONS:
Device: MynxGrip — Vascular Closure
  Arms: MynxGrip
Other: Manual compression — Manual compression is a commonly used method to achieve hemostasis of femoral artery
  Arms: Manual compression

SUMMARY:
To evaluate the safety and effectiveness of MynxGrip, in hemostasis of common femoral artery puncture site, compared with manual compression hemostasis in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F or 7F procedural sheath.

DETAILED DESCRIPTION:
Effectiveness: to superiority to the control group in time to hemostasis. Comparison of time to ambulation, procedure success rate, length of stay in hospital, device success rate.

Safety-Major/Minor complication rate, adverse events, SAEs as compared to control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age;
2. Patients who are able and willing to sign the informed consent form;
3. Patients who agree to follow all study visits and procedures;
4. Patients who plan to receive the diagnostic or interventional endovascular procedures via percutaneous common femoral artery puncture; 5) Patients who are able to walk, as judged by the investigators.

Exclusion Criteria:

1. Patients are proved to have clinically significant peripheral vascular disease according to any of the following situations:

   1. Patients showing severe claudication after walking less than 200 meters,
   2. No palpable pulse on the patients' affected limbs,
   3. Patients having received surgical procedures involving the ipsilateral common femoral artery
   4. Patients having received percutaneous transluminal angioplasty (PTA), stent placement, or vascular graft in the ipsilateral common femoral artery;
2. Patients with morbid obesity (BMI > 40 kg/m2);
3. Patients with a myocardial infarction (MI) with acute elevated ST segment ≤24 hours prior to procedure;
4. Patients with the prior procedure in the ipsilateral common femoral artery ≤30 days;
5. Patients having received ipsilateral vascular closure device;
6. Patients with bleeding disorders such as thrombocytopenia (platelet count < 100,000/ mm3), hemophilia, von Willebrand disease or severe anemia (Hgb < 10 g/dL, Hct < 30%);
7. Patients with documented INR > 1.5 or patients currently receiving glycoprotein IIb/IIIa platelet inhibitors;
8. Patients with symptoms of local infection or inflammation in the groin;
9. Patients who are participating in any other clinical studies on drugs or medical devices at the same time;
10. Patients who are pregnant or in lactation;
11. Patients with known allergy to contrast medium;
12. Patients with known allergy to polyethylene glycol;
13. Patients with treated but still uncontrolled hypertension (systolic pressure>180 mmHg or diastolic pressure>110 mmHg);
14. Patients with known autoimmune diseases;
15. Patients who are receiving long-term corticosteroid therapy;
16. Patients with expected life of less than 30 days;
17. Patients with unilateral or bilateral lower-extremity amputation;
18. Patients who can't walk 6 meters (20 steps) without a support for any reason;
19. Patients requiring prolonged length of stay [For example, the patient will receive the coronary artery bypass grafting (CABG) or the patient plans to receive the CABG ≤30 days after the surgery];
20. Patients with mental disorders and cognitive impairment;
21. Patients have participated into this study before; Intra-operative exclusion criteria;
22. Patients with treated but still uncontrolled hypertension (systolic pressure>180 mmHg or diastolic pressure>110 mmHg);
23. Patients implanted with a balloon pump inside the aorta;
24. Patients whose common femoral artery is too thin (<5 mm in diameter);
25. Patients with obviously fibrotic, calcified, or >50% stenotic femoral artery;
26. Patients having received puncture at other artery than the common femoral artery;
27. Patients having received antegrade puncture;
28. Patients having received arterial puncture at a number of different sites or who are suspected to have received posterior femoral arterial wall puncture;
29. Patients implanted with ipsilateral venous sheath;
30. Surgical findings or complications which the investigators consider may interfere with the patients' participation into the study (For example, the sheath deployment is difficult due to the scar, tortuous vessels, or use of the sheath with the other sizes than 5 Fr, 6 Fr or 7 Fr, or the sheath with the total length of >15.7 cm);
31. Patients with preexisting hematoma, intraluminal thrombus, pseudoaneurysm, AV Fistula or any type of dissection;
32. Patients requiring prolonged length of stay [For example, the patient will receive the coronary artery bypass grafting (CABG) or the patient plans to receive the CABG ≤30 days after the surgery];
33. Patients who are included in another drug or medical device study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | Intraoperatively
  To evaluate whether the time to hemostasis for the puncture site of common femoral artery of the subjects in the MynxGrip group is superior to the control group. Determined using the following formula where time is measured in minutes. H0: ttest - tcontrol ≥ -5，H1: ttest - tcontrol < -5

SECONDARY OUTCOMES:
Time to ambulation | At time of procedure through discharge (up to 3 days post procedure)
  Compare whether there are statistical differences between the test and control group in the time to ambulation measured in hours and determined using a t-test analysis
Length of hospital stay | Up to 5 days post procedure
  Compare whether there are statistical differences between the test and control group in the length of the hospital stay measured in hours and using a t-test analysis.
Procedure Success Rate | Intraoperatively
  Chi-squared Test or Fisher's Exact Test is used, according to the distribution characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Miao Zhongrong, MD, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University
Locations (1):
- Beijing Tiantan Hospital Capitol Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No